CLINICAL TRIAL: NCT05792930
Title: Developing an Integrated Psychotherapy With Cognitive-behavioral Therapy and Biofeedback Therapy for Somatic Symptom Disorder: a Randomized Controlled Trial
Brief Title: Developing an Integrated Psychotherapy With Cognitive-behavioral Therapy and Biofeedback Therapy for Somatic Symptom Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202209093RIND
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Somatic Symptom Disorder
Keywords: somatic symptom disorder; cognitive behavioral therapy; biofeedback therapy; somatic distress; health anxiety
MeSH Terms: interventions — Cognitive Behavioral Therapy; Biofeedback, Psychology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive cognitive-behavioral therapy (CBT) and biofeedback therapy.
  Interventions: Behavioral: cognitive-behavioral therapy and biofeedback therapy
- Control Group (No Intervention): The design of control group is waiting list control; their data will be collected without intervention during the observation period. After the observation period, psychotherapy (CBT and biofeedback, the same as intervention) will be arranged.

INTERVENTIONS:
Behavioral: cognitive-behavioral therapy and biofeedback therapy — Complete eight sessions of cognitive-behavioral therapy and biofeedback therapy within three months.
  Arms: Experimental Group

SUMMARY:
This research program is aimed to develop a integrative psychotherapy (including CBT and biofeedback therapy) and to examine its efficacy on treatment of somatic symptom disorder. The study design is a randomized controlled trial with waiting list control. Scores of Patient Health Questionniare-15 and Health Anxiety Questionnaire are the primary endpoints.

DETAILED DESCRIPTION:
Somatic symptom disorder (SSD) is a psychiatric disorder featured with somatic distress and related psychological phenomena. In the past several years, our research team has investigated several aspects of SSD, including psychopathology, epidemiology, mechanism, and diagnostic biomarkers. But the aspect about treatment on SSD has not been comprehensively explored.

In literature, the treatment of SSD can be separated into physical and psychological approaches. The physical approach includes pharmacotherapy and magnetic/electrical neuromodulation. Among several types of psychotherapies, cognitive behavioral therapy (CBT) has the most evidence. Previous studies have disclosed SSD patients to have following cognitive or behavioral features: selective attention on somatic distress; memory bias on the severe health conditions; all-or-none cognition about health; organic attribution style; catastrophizing cognitive pattern about health; high motivation of concerning issues about health; inadequate reassurance-seeking behavior; the assumption about the connection between rest and somatic distress, etc.

Biofeedback therapy works by measuring several biological signals related with stress and relaxation (such as heart rate, skin conductance, electromyography, electroencephalography, and finger temperature); feedback of these signals to the subjects can help them more clearly understand the association between their behavior/cognition and relaxation. Biofeedback therapy has been extensively applied in the psychosomatic field.

This research program is aimed to develop a integrative psychotherapy (including CBT and biofeedback therapy) and to examine its efficacy. The study design is a randomized controlled trial with waiting list control. Scores of Patient Health Questionniare-15 (PHQ-15) and Health Anxiety Questionnaire (HAQ) are the primary endpoints; the changes of other psychological and biological measurements are viewed as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patient with somatic symptom disorder (confirmed by psychiatrists)

Exclusion Criteria:

* The age is younger than 20 or older than 70 years
* Having psychotic symptoms or cognitive impairment
* Having a potentially lethal illness
* Cannot read the questionnaires by oneself

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Scores of Patient Health Questionnaire-15 (PHQ-15) | Week 12 (comparing with the data in week 0)
  Measurement of somatic distress. Score range is 0 to 30; higher score means more severe somatic distress
Scores of Health Anxiety Questionnaire (HAQ) | Week 12 (comparing with the data in week 0)
  Measurement of health anxiety. Score range is 0 to 63; higher score means more severe health anxiety

SECONDARY OUTCOMES:
Scores of Beck Depression Inventory-II (BDI-II) | Week 12 (comparing with the data in week 0)
  Measurement of depression. Score range is 0 to 63; higher score means more severe depression
Scores of Beck Anxiety Inventory (BAI) | Week 12 (comparing with the data in week 0)
  Measurement of anxiety. Score range is 0 to 63; higher score means more severe anxiety
Scores of Cognitions About Body and Health Questionnaire (CABAH) | Week 12 (comparing with the data in week 0)
  Measurement of cognitions about health. Score range is 0 to 117; higher score means more severe cognitive distortion about health
Heart rate variability | Week 12 (comparing with the data in week 0)
  Measurement of parasympathetic activity
Skin conductance | Week 12 (comparing with the data in week 0)
  Measurement of sympathetic activity

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Lieh Huang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital Yunlin Branch, Yunlin, Taiwan